CLINICAL TRIAL: NCT05440630
Title: Efficacy and Safety of Probiotic Strain Bifidobacterium Animalis Subsp. Lactis CECT 8145 Probiotic in the Reduction of Abdominal/Visceral Fat in Overweight and Obese Patients: Double-blind, Randomised, Placebo-controlled Trial
Brief Title: Study of Efficacy of a Probiotic and Postbiotic in Overweight and Obese Individuals
Acronym: Obelix
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to ship investigational product to trial site.
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: Nois de México (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCTB202015
Record Dates: First submitted 2022-06-16; First posted 2022-07-01 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic (Experimental): Participants in this arm will receive a daily dose of 1x10^10 Colony Forming Unit (CFU) of a single strain probiotic (live bacteria) for 16 weeks.
  Interventions: Dietary Supplement: Probiotics
- Postbiotic (Experimental): Participants in this arm will receive a daily dose of 1x10^10 Colony Forming Unit (CFU) of a single strain probiotic (Heat treated bacteria) for 16 weeks.
  Interventions: Dietary Supplement: Postbiotic
- Placebo (Placebo Comparator): Participants in this arm will receive an equivalent placebo for 16 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Participants in this arm will receive a daily dose of 1x10^10 Colony Forming Unit (CFU) of a single strain probiotic (live bacteria) for 16 weeks.
  Arms: Probiotic
Dietary Supplement: Postbiotic — Participants in this arm will receive a daily dose of 1x10^10 Colony Forming Unit (CFU) of a single strain postbiotic (Heat treated bacteria) for 16 weeks.
  Arms: Postbiotic
Dietary Supplement: Placebo — Participants in this arm will receive an equivalent placebo for 16 weeks.
  Arms: Placebo

SUMMARY:
The study's main objective is to investigate the effect of a probiotic (live bacteria), postbiotic (heat-treated bacteria) on obesity parameters.

DETAILED DESCRIPTION:
Investigation of the efficacy of probiotics as adjuvant in the management of overweight and obesity. Specifically, in the reduction of abdominal/visceral adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects from 18 to 65 years old.

Established diagnosis of overweight (BMI ≥ 25 and up to 34.9)

Waist circumference ≥ 102 cm for men

Waist circumference ≥ 88 cm for women

Signature of the informed consent letter.

Agreement to comply with the protocol and study restrictions

Exclusion Criteria:

Diagnosed and pharmacologically-treated type 1 or type 2 diabetes

Subjects with serious autoimmune disease, cardiovascular disease, liver dysfunction/disease, kidney dysfunction/disease or chronic disease

Immunosuppression or ongoing therapy causing immunosuppression

Pharmacologically-treated (medication/supplements) hypertension or dyslipidaemia

Subjects consuming antibiotics in the previous 2 months

Subjects consuming probiotics and prebiotics at least 1 month prior to inclusion in the study or during the intervention period.

History of chronic active inflammatory disorders

History of bariatric surgery

History of any chronic gastrointestinal disease (e.g. IBD).

Known hypersensitivity to any ingredients in the active or placebo products.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in abdominal/visceral fat area | 0 week to 16 week
  Difference in abdominal visceral fat area on MRI from baseline (V1) to 4 months of product intake (V4) within and between groups.

SECONDARY OUTCOMES:
Change in abdominal subcutaneous fat area | 0 week to 16 week
  Difference in abdominal subcutaneous fat area on MRI from baseline (V1) to 4 months of product intake (V4) within and between groups.
Change in body composition | 0 week to 16 week
  Difference in total body fat mass (kg) from baseline to 4 months of product intake within and between groups (relative and absolute, measured by bioelectrical impedance at V1 and V4).
Change in body weight | week 0, week 4, week 8, week 16
  Body weight change (percent and kg) at all visits - difference within and between groups.
Change in BMI | week 0, week 4, week 8, week 16
  BMI change (units and percent) at all visits - difference within and between groups.
Change in waist circumference | week 0, week 4, week 8, week 16
  Change in waist circumference (all visits V1-4)
Change in hip circumference | week 0, week 4, week 8, week 16
  Change in hip circumference at all visits difference within and between groups (absolute and relative)
Change in lipid profile | week 0, week 16
  Change in total cholesterol, triglycerides, LDL, VLDL and HDL (mg/dL) (baseline and 4 months)
Change in systolic and diastolic blood pressure | week 0, week 4, week 8, week 16
  Change in systolic and diastolic blood pressure (mmHg)
Changes in glucose profile | week 0, week 16
  Change in HOMA-IR (fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5)
Change in cortisol levels | week 0, week 16
  Change in cortisol levels (nmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Joshue Covarrubia Esquer, Dr, Principal Investigator — NOIS DE MEXICO S.A. DE C.V.
Locations (1):
- Nois de Mexico S.A. de C.V., Guadalajara, Mexico

IPD SHARING:
Plan to Share IPD: No